CLINICAL TRIAL: NCT06677489
Title: Prognostic Modeling of Heart Failure Risk in a Large-Scale Asian Cohort With Chronic Kidney Disease: The CKD-Heart Study
Brief Title: CKD-Heart: Heart Failure Prediction in Asian CKD Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chung-Lieh Hung, • Director of Ultrasound Imaging and Telemedicine, Cardiovascular Center, Mackay Memorial Hospital • Director of the Department of Heart Failure and Imaging Medicine, Cardiovascular Center, Mackay Memorial Hospital, Mackay Memorial Hospital
Other Study IDs: 23MMHIS240e
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease(CKD)
Keywords: cardiovascular disease; biomarkers; chronic kidney disease; heart failure; echocardiogram
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Among patients with known chronic kidney disease (CKD) who are free from diagnosed heart failure (HF), some may be classified as stage A-B HF based on the contemporary 2022 ACC/AHA Guideline for Heart Failure Classification. Several key clinical features and risk factors have been shown to serve as predictors for future HF development. Importantly, compared to white populations, Asians may present with distinct HF risks even when exhibiting the same conventional clinical risk factors for CKD.

Our current study aimed to explore the clinical predictors of HF and adverse cardiovascular events among CKD patients in a pre-clinical HF stage (Stage A-B) within a large ethnic Asian population. We further investigated whether baseline characteristics from echocardiography, ECG, and urine protein measurements could provide additional prognostic insights on future events. Addressing this knowledge gap for such a population may facilitate early identification and timely interventions for CKD patients of Asian ethnicity in the early stages of the disease.

DETAILED DESCRIPTION:
1.1 Background and rationale for conducting this study

Patients with chronic kidney disease (CKD), a clinical scenario closely associated with multiple co-morbid conditions (e.g., hypertension, diabetes, and coronary artery diseases), are less likely to receive guideline-directed foundational medical therapy due to clinical concerns about hyperkalemia and hypotension, and are thereby prone to the development of heart failure (HF). In this regard, early identification and prevention of HF is important (1). To date, N-terminal pro-brain natriuretic peptide (NT-pro-BNP) has been shown to be a powerful clinical predictor of HF, though its clinical utilization is easily affected by renal insufficiency, thus limiting its use in these patients (2).

1.2 Rationale for study design, doses and control groups

Overall rationale and study population:

Recent studies have shown improvement in cardiovascular outcomes, particularly in HF, and renal protective effects of SGLT2 inhibitors (3). Early identification of HF among CKD patients in a pre-clinical HF stage may allow appropriate pharmacological interventions as early as possible to reduce future HF burden. Yet, data regarding the exact clinical characteristics and risk stratification for HF diagnosis in CKD subjects that may benefit from interventions remain largely unexplored.

Whether the use of several key baseline clinical risk factors, including baseline eGFR (using MDRD or CKD-EPI formula), Urine albumin to creatinine ratio (UACR), serum biomarkers (NT-proBNP, hs-CRP, or hs-TNI), either combined or alone, among CKD ethnic Asians at a pre-clinical HF stage (without prevalent HF) or at a time point where early therapeutic intervention may be beneficial for such patients in daily practice remains to be determined from large-scale real-world datasets. We further aim to explore the clinical cut-off of NT-proBNP in identifying incident HF in CKD patients applicable to ethnic Asians based on a large-scale CKD population.

Prior evidence: 51% of heart failure patients have an eGFR <60 mL/min/1.73 m2 and 11% have an eGFR <30 mL/min/1.73 m2. Increasing mortality was found as kidney function decreased, regardless of the presence of diabetes, age, hemoglobin levels, New York Heart Association (NYHA) class, and duration of heart failure (4). Kidney dysfunction is not only correlated with short-term and long-term outcomes in patients with heart failure but is also a predictor for the risk of heart failure (5).

Objectives:

Use several key clinical risks, for example, Framingham heart study risk factors and variables collected in the CRIC study (6), to early identify HF events among CKD patients free from prevalent HF; Explore the clinical cut-off of NT-proBNP in identifying HF in CKD patients in Taiwan.

Unique aspects: The risk factors identified by the CRIC (Chronic Renal Insufficiency Cohort) study are not commonly used for clinical daily practice, for example, insulin resistance, inflammation, and hsTnI (6, 7). We would like to use CRIC clinical scores including clinical demographics (e.g., age, blood pressure, smoking, and medical comorbidities), echo-based parameters (e.g., LVM, LVEF), biomarkers (e.g., hsTnT and NT-proBNP), and renal profiles (eGFR and UACR), to identify high-risk HF in CKD patients. Besides, the cut-offs of eGFR/UACR/hs-TnI/NT-proBNP to identify HF among large-scale Asian CKD patients are not clear.

Expected data:

Identify several key clinical risk factors that are easy to obtain for clinical practice to early identify HF in CKD among a large-scale Asian cohort.

Find out the optimal cutoff of eGFR (using different formulas, such as MDRD or CKD-EPI) and UACR in predicting HF incidence in CKD patients.

1.3 Benefit/risk and ethical assessment

Benefit:

Identification of HF predictors among CKD patients in pre-clinical HF stage (Stage A-B) prior to overt clinical HF.

Besides, eGFR/UACR, hs-TnI/NT-proBNP checkup as routine to identify HF risk may not be generalizable in asymptomatic CKD patients.

Risk:

Not applicable

Ethical assessment:

This protocol will be reviewed by IRB.

1.4 Study Design

Study group:

Retrospective study: Pooled 9000-10000 CKD patients from Mackay Memorial Hospital (2-center pooled data) Data collection range: retrospective, starting from 2011-2020 Data collection timeline: half a year

Several clinical risk factors and NT-ProBNP level at baseline and subsequent vascular events up to 5 years in a retrospective manner will be collected. Associations of these clinical risks with the development of HF and vascular events will be established.

Data collection content:

* Framingham risk factors and CRIC study-based clinical variables including age, HDL-C, total cholesterol, blood pressure, HbA1c, smoking habit, IL-6, TNF-α, insulin resistance, anemia, albuminuria or ACR (urine albumin/creatinine ratio), and hs-TnI will also be collected if available.
* Data regarding conventional echocardiography parameters for indexed LV mass and LV ejection fraction (LVEF) will also be collected if available.
* Diabetes and dialysis duration will be collected if available.
* Long-term used (i.e., with ≥ 6 months treatment duration) medications that may affect renal function and heart function will be collected (ACEi/ARB, MRA, ARNI, SGLT2i, diuretic, TZD, GLP-1 RA, and NSAID)

Follow-up: clinical events (vascular events including stroke, myocardial infarction, unstable angina or elective PCI, atrial fibrillation (AF), atrial flutter (AFL), heart failure (HF), and any cause of death event) up to 5 years in a retrospective manner following the index date of data collection for any individual.

Echocardiography Sub-study:

* Echocardiography features in symptom-free CKD of ethnic Asians
* Prevalence and prognostic utilization of diastolic dysfunction in symptom-free CKD among ethnic Asians

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CKD (an estimated glomerular filtration rate (eGFR) of less than 60 mL/min/1.73 m², persisting for 3 months or more)
* Age ≥ 20 years
* Free at baseline of diagnosed HF
* Baseline patient-level clinical data available

Exclusion Criteria:

* Known HF hospitalization history
* Known impaired LV systolic function (LVEF<40%) by any imaging modality
* Any terminal disease other than CKD lowering the patient's life expectancy to less than two years
* eGFR ≥ 60ml/min/1.73m2

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study group:
  Retrospective study: Pooled data from 9000-10000 CKD patients at Mackay Memorial Hospital Data collection range: retrospective data collection from 2011 to 2020
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incident heart failure (HF), Cardiovascular death (CV Death) and All-cause death | From enrollment to the end of observation for at least 5 years

SECONDARY OUTCOMES:
1. Non-fatal cardiovascular events or CV Death (MACE), Atrial fibrillation (AF)/Atrial flutter (AFL) related hospitalization; 2. Echocardiography defined structural and functional abnormalities. | From enrollment to the end of observation for at least 5 years
  2. Echocardiography defined structural and functional abnormalities including: A. Cardiac structures IVS, mm LV posterior wall, mm LVIDd, mm LVEDV, ml LVESV, ml RWT, mm LV mass, g LV mass index, g/m2.7 B.Diastolic function DT, ms IVRT, ms E, cm/s e' (lateral), cm/s E/e' (lateral) A, cm/s C. Systolic function LVEF, % GCS , % LVSRe, s-1 LVSRa, s-1 LVSRs, s-1 Torsion, °/cm

CONTACTS AND LOCATIONS:
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No